CLINICAL TRIAL: NCT06678022
Title: Use of Unmanned Air Vehicles (Medical Drones) to Overcome Geographical Barriers to Delivery of Anti-Retrovical Samples: A Cluster Randomised Trial in Kalangala District, Uganda
Brief Title: Use of Unmanned Air Vehicles (Medical Drones) to Overcome Geographical Barriers to Delivery of Anti-Retroviral Therapy and Biological Samples
Acronym: MRC-DRONES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Medical Research Council (Other Government); United Kingdom Research and Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAKSPHREC 007/2020; MRC AGHRB - MR/Y019717/1 (Other Grant/Funding Number: MRC-UKRI (MRC and the International Science Partnerships Fund (ISPF)))
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: HIV; Viral Load
Keywords: virological suppression; Fisher Folk; Cluster Randomised Trial; medical drones

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial using a non-inferiority design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Delivery of ART by fixed wing drones to landing sites
  Interventions: Device: Fixed Wing drones
- Control arm (Active Comparator): Usual ART delivery to landing sites
  Interventions: Device: No Drone delivery

INTERVENTIONS:
Device: No Drone delivery — Usual ART delivery to landing sites
  Arms: Control arm
Device: Fixed Wing drones — Last Mile fixed wing drone delivery
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to learn if the intervention of delivery of antiretroviral drugs by medical drones can improve virological suppression in a fisherfolk community population living with HIV in the islands of Kalangala District, Uganda. The main question it aims to answer is:

Can delivery of anti-retroviral therapy (ART) by unmanned aerial vehicles (medical drones) to people living with HIV (PLHIV) improve virological outcomes compared to the standard of care (SOC) in an underserved population? Primary hypothesis: The investigators hypothesize that using drones will increase viral suppression in those receiving the intervention as compared to the control or outcome measure one-will be the proportion of PLHIV with undetectable HIV viral load in the intervention (drones) versus SOC arm at 12 months.

If there is a comparison group: Researchers will compare [Medical Drones delivery group] to see total cost of 12 months medication delivery to people living with HIV (PLHIV) in the intervention as compared to standard of care (SOC) arm.

Proportion PLHIV with an undetectable viral load at 6, 18 and 24 months in intervention Rates of retention in care of PLHIV at 6,12, 18 and 24 months in intervention as compared to SOC arm

* Participants will be seen every 6 months for 24 months
* They will have blood draws for viral load tests
* They will complete interviewer administered questionnaires
* The intervention is last-mile delivery of ART by drones to landing sites

DETAILED DESCRIPTION:
The Investigators will undertake a cluster randomised trial of the efficacy of medical drone use by randomization of health facilities and their associated landing sites in Kalangala District. There are 64 landing sites and 18 health facilities. The unit of radomisation will be the landing site, so that all persons at one landing site will receive the drone delivery or boat delivery, facility pick-up. This will avoid contamination of drone delivery by sharing of ART between people getting drone and boat or other modes of deliveries. Bias in this situation will be managed by stratifying the landing sites by distance from drone operations base (a proxy of delivery cost), and number of differentiated service delivery (DSD) groups. Bias in gender and age will be managed at selection of members in DSD groups. We will also undertake a cost effectiveness analysis, carbon analysis and process evaluation. A qualitative study will assess acceptability and additional use cases

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) living with HIV
* Emancipated minor (15-17 years) who is living with HIV
* Receiving antiretroviral therapy in Kalangala District
* Be a resident in Kalangala district for at least the preceding 6-12 months
* Willing to stay for a minimum next 24 months
* Willing to disclose HIV status to an expert peer or village health team member.
* Willing to join discentralised Service Delivery model groups

Exclusion Criteria:

* Potential participants below 15 years with care providers not receiving care from DSD.
* No active opportunistic infection (including but not limited to TB) in health centre records or self-report or suspected by the study team at enrolment (will be referred back to health facility for investigations and can be enrolled if no infection confirmed).
* Patients with mental illness or any other medical condition that compromises decision making process (as determined by medical records at facility and direct questioning to participant)
* Any other clinical condition that, in the opinion of the site investigator, would make the participant unsuitable for the study or unable to comply with dosing requirements.
* For stage three, participants residing in areas that took part in stage 2 drone delivery eg Bufumira island

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1086 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
primary endpoint is the proportion of participants with HIV RNA viral load < 200 copies/mL at 12 months | 12 months
  Analysis of the primary endpoint shall be done on modified intention-to-treat population, mITT (i.e. includes all participants randomized, and received at-least one dose of treatment). We shall use log-binomial/Poisson mixed effects regression model to compare proportion of PLHIV with an undetectable HIV viral load (i.e. <200 copies/mL) at month 12 between the two arms

SECONDARY OUTCOMES:
Intermediate and final 12-month retention in care in those receiving ART via drone compared to control population | 12 months
  Retention in care defined as participant with a facility or ART encounter for > 90 days after the last missed scheduled ART collection
proportion of viral load > 200 copies/mL at 24 | 24 months
  Proportions be summarised by the treatment arms and compared used Pearson Chi-square test.

CONTACTS AND LOCATIONS:
Locations (2):
- Uganda (2):
  - Bwendero Health Centre, Kalangala, Ssese
  - Mugoye health Centre III, Kalangala, Ssese

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the trial will be shared at the end of the project after manuscript have been completed.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Start dates 2027 No limit/end
Access Criteria: All interested researchers, policy makers, participants. Can access the data sets, clinical reports, monitoring reports, DSMB reports
URL: https://theacademy.co.ug/medical-drones-project

REFERENCES:
- See also: Related Info — https://theacademy.co.ug/medical-drones-project/